CLINICAL TRIAL: NCT03375944
Title: The Use of Modern Telemedicine Technologies in an Innovative Program of Optimal Cardiac Rehabilitation in Patients After Completed Myocardial Revascularization
Brief Title: Utilisation of Telemedicine in Optimal Cardiac Rehabilitation Program in Patients After Myocardial Revascularization
Acronym: RESTORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pawel Buszman (Other)
Responsible Party: Sponsor-Investigator, Pawel Buszman, Chief Executive Officer, American Heart of Poland
Organization: American Heart of Poland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RESTORE2015
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Coronary Artery Disease With Myocardial Infarction
Keywords: Cardiac tele-rehabilitation, Myocardial revascularization
MeSH Terms: conditions — Coronary Artery Disease, Autosomal Dominant, 1 | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Cardiac supervision
- study group (Other): Cardiac supervision and rehabilitation
  Interventions: Other: Rehabilitation

INTERVENTIONS:
Other: Rehabilitation — The purpose of this work package is to evaluate short- and long-term clinical effects of optimal, continuous and regularly controlled tele-rehabilitation, which is based on exercise training, intensive dietary and educational program focused on lifestyle and risk factors modification. The main expectations of OCR is to normalize annual mortality to the level of the low risk "healthy" population.
  Arms: study group

SUMMARY:
Although clinical data demonstrate advantages of combining complete revascularization with optimal cardiac rehabilitation (CR) less than one-third of patients in European countries participate in cardiac rehabilitation programs. Therefore, in cooperation with Polish leaders in cardiovascular medicine, rehabilitation and medical software design we aim to introduce and evaluate the system of optimal cardiac telerehabilitation in addition to optimal treatment of coronary artery disease.

DETAILED DESCRIPTION:
Although clinical data demonstrate advantages of combining complete revascularization with optimal cardiac rehabilitation (OCR) less than one-third of patients in European countries participate in cardiac rehabilitation programs.

In addition, the major limitations of current CR programs are their short duration without long-term follow-up, lack of appropriate clinical and functional monitoring, and structural problems including geographic misdistribution of available programs. Therefore, in cooperation with Polish leaders in cardiovascular medicine, rehabilitation and medical software design we aim to introduce and evaluate the system of optimal cardiac telerehabilitation in addition to optimal treatment of coronary artery disease. Primarily, the telerehabilitation system will be designed and developed. Secondly, coordinating center will be build and technical tests will be performed in order to evaluate its integrity with telerehabilitation system. Thirdly, the whole system will be validated in clinical settings on patients' population with coronary artery disease and completed revascularization. Finally, procedural steps will be executed in order to prepare the whole system of optimal cardiac telerehabilitation for implementation.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 and below 70
* completed revascularization in patients with stable or unstable angina or after myocardial infarction without ST-segment elevation (NSTEMI)
* in patients with suspected myocardial scars, MRI will be recommended to confirm myocardial viability.
* eligibility to participate in a program of early cardiac rehabilitation
* signed informed consent form
* the ability to use telerehabilitation system

Exclusion Criteria:

* acute myocardial infarction with ST segment elevation/new onset of left bundle branch block (LBBB),
* suboptimal (not completed) revascularisation
* ejection fraction <40%.
* acute heart failure (Killip IV) at the time of admission to the hospital
* dual antiplatelet therapy can not be maintained for 1 year after PCI
* haemorrhagic stroke in the past
* ischemic stroke or transient ischemia in previous 6 weeks
* platelet count <100,000 / mm3
* chronic renal failure with creatinine clearance <30ml / min / 1.73m2
* planned surgery
* pregnancy or planned pregnancies
* expected life expectancy less than 3 years after enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 12 months
  The primary objective of the study is to compare the all cause mortality between the control and the study group during the annual follow-up.
All cause mortality | 9 months
  The primary objective of the study is to compare the all cause mortality between the control and the study group during the 9-month follow-up.

SECONDARY OUTCOMES:
Rate of major adverse coronary and cerebrovascular events (MACCE) | 9 months and 1 year
  MACCE defined as either: any cause death, repeat revascularization, myocardial infarction and stroke at 1 year follow-up,
rate of target vessel failure (TVF) | 9 months and 1 year
  TVF defined as composite of death, myocardial infarction or target vessel revascularization
cardiac death | 9 months and 1 year
  all cause and cardiac death will be recorded
Length of hospital stay | up to 9 months and 1 year
  total hospital length will be recorded
Regression, stabilisation or progression of atherosclerotic plaques | baseline + up to 1 year follow-up
  Measured in coronary arteries with the use of IVUS/NIRS (Intravascular Ultrasound / Near-infrared spectroscopy)
Molecular changes in blood | up to 1 year follow-up
  Multiple molecular parameters will be measured at baseline and at 9-12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Milewski, MD PhD, Principal Investigator — American Heart of Poland
Locations (5):
- Poland (5):
  - Malopolskie Centrum Sercowo-Naczyniowe, Chrzanów, Lesser Poland Voivodeship
  - IV Oddział Kardiologii Inwazyjnej, Elektrostymulacji i Angiologii, Kedzierzyn Kozle, Lower Silesian Voivodeship
  - II Oddział Kardiologiczny, Bielsko-Biala, Upper Silesia
  - III Oddział Kardiologii Inwazyjnej, Angiologii i Elektrokardiologii, Dąbrowa Górnicza, Upper Silesia
  - X Department of Interventional Cardiology, Tychy, Upper Silesia

IPD SHARING:
Plan to Share IPD: No